CLINICAL TRIAL: NCT07298837
Title: The Effect of Turtle Therapy on HbA1c and Self-Efficacy Levels in Diabetes Medication Use in Individuals With Type 2 Diabetes: A Double-Blind Randomized Controlled Study
Brief Title: Turtle Therapy on HbA1c and Self-Efficacy Levels With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RCS04072024
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus; Pet-Human Bonding
Keywords: Hemoglobin A1c Test; Pet Therapy; Self-efficacy; Turtle Therapy; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Human-Animal Bond | interventions — Animal Assisted Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live Turtle Group (Experimental): Before starting the study, a nurse who was unaware of the study details (to prevent bias) administered the "Structured Patient Information Form" and "Diabetes Medication Self-Efficacy Scale", and the "hemoglobin A1c " value measured immediately before the study began was recorded. At the end of the three-month pet therapy period, the same nurse administered the "Diabetes Medication Self-Efficacy Scale" test, and the physician recorded the "hemoglobin A1c" value result as requested. During this process, patients continued their routine Type 2 Diyabetus Mellitus treatment.
  Interventions: Behavioral: Live Turtle Therapy (Pet therapy)
- Video Turtle Group (Experimental): Before starting the study, a nurse who was unaware of the study details (to prevent bias) administered the "Structured Patient Information Form" and "Diabetes Medication Self-Efficacy Scale", and the "hemoglobin A1c" value result measured immediately before the study began was recorded.In addition, at the end of the three-month pet therapy period, the same nurse administered the "Diabetes Medication Self-Efficacy Scale" and the physician recorded the "hemoglobin A1c" value result requested. During this process, patients continued their routine Type 2 Diyabetus Mellitus treatment.
  Interventions: Behavioral: Video Turtle Therapy (Pet therapy)
- Control Group (No Intervention): A nurse who was unaware of the study details prior to its commencement (to prevent bias) administered the "Structured Patient Information Form" and "Diabetes Medication Self-Efficacy Scale", and the "hemoglobin A1c" value result obtained immediately before the study began was recorded. No intervention was performed on these patients. Patients only continued their routine Type 2 Diyabetus Mellitus treatments. In addition, "Diabetes Medication Self-Efficacy Scale" was administered to patients at the end of the three-month period, and the "hemoglobin A1c" value requested by the physician was recorded.

INTERVENTIONS:
Behavioral: Live Turtle Therapy (Pet therapy) — The individuals were asked to take on the responsibility of caring for the turtles. The patients in this group were given one turtle and the necessary materials (aquarium, food, aquarium sand, etc.) for 12 weeks. Within this scope, patients fed the turtles twice a day, once in the morning (08:00) and once in the evening (20:00), and changed the water in the aquarium every two days with water that had been kept at room temperature beforehand. In addition, they were asked to spend 20 minutes a day with the turtle. During the twelve-week (3-month) period in which the individuals took responsibility for turtle care, the "Turtle Monitoring Form" was administered by the executor to evaluate the time spent with the turtle and the implementation of practices related to how they performed turtle care.
  Arms: Live Turtle Group
Behavioral: Video Turtle Therapy (Pet therapy) — In addition, the consultant faculty member provided approximately 15 minutes of face-to-face information to patients regarding watching the turtle videos. Patients in this group were asked to watch documentaries featuring turtle videos for at least 20 minutes a day for twelve weeks. The "Turtle Viewing Form" was administered by the researcher to determine how many minutes per day the individuals watched the turtle videos.
  Arms: Video Turtle Group

SUMMARY:
This study examined the effect of live and video turtle therapy on hemoglobin A1c tests and self-efficacy levels in adults with Type 2 Diabetes Mellitus for the first time using pre-test and post-test methods.

DETAILED DESCRIPTION:
In the international literature reviewed, only two studies reported that pet therapy reduced hemoglobin A1c tests and increased self-efficacy in adolescents with Type 1 Diabetes Mellitus. One study examined the use of live fish (repeated care behaviors during pet care, such as feeding twice a day and cleaning the aquarium). In the other study, adolescents who owned different types of pets (dogs, cats, birds, fish, reptiles, amphibians, rodents, etc.) were included in the study. In this context, our study will be the first study conducted in individuals with Type 2 Diabetes Mellitus using live and video turtle therapy at the national and international level. With the theoretical clarification of the methodological steps, this study, which has methodological characteristics, is unique in that it compares live animal (turtle) and video animal (turtle video) therapy in individuals with Type 2 Diabetes Mellitus, making it a pet therapy study conducted both nationally and internationally in both turtles and individuals with Type 2 Diabetes Mellitus. Within the scope of all this information, this study examined the effect of live and video turtle therapy on hemoglobin A1c and self-efficacy levels in adults with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Agreement to participate in the study,
* Being literate,
* Being able to communicate verbally,
* No vision, hearing, or speech impairments,
* Agreeing to adopt and care for a turtle (turtle group),
* Ownership of a smartphone, tablet, or computer (video turtle group),
* Having been diagnosed with T2DM and having been receiving DM treatment for at least 6 months,
* HbA1c >7%.

Exclusion Criteria:

* Refusal to participate in the study,
* Not having T2DM,
* Having received DM treatment for less than 6 months,
* Having a psychiatric disorder diagnosed by a psychiatrist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 week
  Hemoglobin A1c is a clinically useful index of average blood glucose levels over the past 120 days (average red blood cell lifespan). It most accurately reflects glycemic control over the past 2-3 months.
  Hemoglobin A1c was measured twice, before and after the study.
Diabetes Medication Self-Efficacy Scale | 12 week
  Diabetes Medication Self-Efficacy Scale was developed by Sleath and colleagues (2016) to assess self-efficacy in overcoming barriers to diabetes medication use. Its Turkish validity and reliability were established by Kavuran & Türkoğlu (2022) using a 19-item, 3-point Likert-type scale. The scale consists of three subscales: "Requirement" (items 1-4), "Busyness" (items 5-9), and "Worry" (items 10-19). The scale scores range from 19 (low self-efficacy) to 57 (high self-efficacy).
  Diabetes Medication Self-Efficacy Scale was measured twice, before and after the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I'll decide later